CLINICAL TRIAL: NCT03587376
Title: Characterization of T-Cell Response in Subjects Previously Treated With JNJ-54861911 (Atabecestat)
Brief Title: Characterization of T-Cell Response in Participants Previously Treated With JNJ-54861911 (Atabecestat)
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CR108462; 54861911ALZ0002 (Other: Janssen Research & Development, LLC); 2018-000403-17 (EudraCT Number: European Medicines Agency (EudraCT))
Record Dates: First submitted 2018-07-04; First posted 2018-07-16 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — atabecestat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants with Elevated Liver Enzymes (Experimental): Blood samples will be collected on Day 1 from participants previously treated with atabecestat and who had elevated liver enzymes while on atabecestat.
  Interventions: Drug: Atabecestat
- Participants Without Elevated Liver Enzymes (Active Comparator): Blood samples will be collected on Day 1 from participants who completed at least 3 months of dosing with atabecestat and who did not have the elevated liver enzymes (adverse event) while on atabecestat.
  Interventions: Drug: Atabecestat

INTERVENTIONS:
Drug: Atabecestat — Blood samples will be collected from participants previously treated with atabecestat.
  Other Names: JNJ-54861911

SUMMARY:
The purpose of this study is to determine T-cell mediated inflammatory immune response in some participants previously exposed to atabecestat.

DETAILED DESCRIPTION:
This is an exploratory Phase 0 study in participants who previously participated in studies (54861911ALZ2002 [NCT02260674], 54861911ALZ2003 [NCT02569398], or 54861911ALZ2004 [NCT02406027]) with atabecestat. In this study, participants will only have blood drawn. The primary hypotheses for this study is that adverse event of elevated liver enzymes observed in some participants is caused by a T-cell dependent inflammatory response. Participants will be monitored for adverse events and will be called 1 day after the blood draw to assess for any adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Participant who received and discontinued atabecestat in one of the following prior trials (54861911ALZ2002, 54861911ALZ2003, or 54861911ALZ2004)
* Must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Willing and able to adhere to the prohibitions and restrictions specified for this study

Exclusion Criteria:

* Anemic based on the last blood draw in the prior atabecestat trial
* Donated more than (>) 450 milliliter (mL) of blood in the past 3 months
* Currently participating in an atabecestat study (54861911ALZ2002, 54861911ALZ2003, or 54861911ALZ2004)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Atabecestat-Specific T-cell Mediated Inflammatory Immune Response | Day 1
  Number of Participants with Atabecestat-Specific T-cell Mediated Inflammatory Immune Response (via cluster of differentiation [CD] 4+ T-cells and CD8+ T-cells) will be determined.

SECONDARY OUTCOMES:
Participants T-cell Receptor (TCR) Sequencing | Day 1
  Participants TCR sequencing will be performed to determine if any particular TCR repertoire is associated with a risk of developing an elevation in liver enzymes following exposure to atabecestat. Participants T-cell receptor repertoire will be sequenced via TCR sequencing techniques.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (5):
- Ziekenhuis Hoge Beuken, Hoboken, Belgium
- Hôpital Fernand Widal, Paris, France
- CTC North GmbH & Co. KG, Hamburg, Germany
- Fundacion Ace, Barcelona, Spain
- Minnesmottagningen, M51, Stockholm, Sweden